CLINICAL TRIAL: NCT02838134
Title: The Effectiveness of Deep Versus Moderate Muscle Relaxation During Laparoscopic Donor Nephrectomy in Enhancing Postoperative Recovery
Brief Title: Deep Versus Moderate Muscle Relaxation During Laparoscopic Donor Nephrectomy in Enhancing Postoperative Recovery
Acronym: RELAX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL58160.091.16
Record Dates: First submitted 2016-06-29; First posted 2016-07-20 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2018-04

CONDITIONS: Neuromuscular Block; Renal Transplant Donor of Left Kidney; Renal Transplant Donor of Right Kidney; Surgery
Keywords: Laparoscopic donor nephrectomy; Early quality of recovery
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Deep Neuromuscular blockade (Experimental): An extra bolus of rocuronium after intubation followed by infusion
  Interventions: Other: Rocuronium
- Group B: Moderate neuromuscular Blockade (Sham Comparator): Moderate neuromuscular Blockade No additional rocuronium after intubation.
  Interventions: Other: No additional Rocuronium

INTERVENTIONS:
Other: Rocuronium — A bolus of 0.7 mg/kg rocuronium is administered just after tracheal intubation and then an infusion of rocuronium (0.3 to 0.4 mg/kg) is started when post-tetanic count (PTC) is more than 0 and titrated towards PTC 1-2.
  Arms: Group A: Deep Neuromuscular blockade
Other: No additional Rocuronium — No additional rocuronium is administered after tracheal intubation.
  Arms: Group B: Moderate neuromuscular Blockade

SUMMARY:
Postoperative recovery after live donor nephrectomy (LDN) is largely determined by the consequences of postoperative pain and analgesia consumptions. The investigators' goal is to establish the relationship between the use of deep neuromuscular blockade (NMB) during laparoscopic donor nephrectomy (LDN) and the early quality of recovery. Therefore, the investigators designed a trial in which patients scheduled for living donor nephrectomy are randomized into a group with deep NMB or moderate NMB. The primary outcome measurement will be the Quality of Recovery-40 questionnaire (overall score) at 48 hours after extubation.

DETAILED DESCRIPTION:
Rationale: Postoperative recovery after live donor nephrectomy (LDN) is largely determined by the consequences of postoperative pain and analgesia consumptions. The use of deep neuromuscular blockade (NMB) has shown to reduce postoperative pain scores after laparoscopic surgery. With this study the investigators will investigate if deep NMB also improves the early quality of recovery after LDN.

Objective: To establish the relationship between the use of deep neuromuscular blockade (NMB) during laparoscopic donor nephrectomy (LDN) - with standard pressure pneumoperitoneum - and the early quality of recovery.

Study design: A multicenter, blinded, randomized controlled trial

Study population: 96 adult patients (18 years or older), scheduled for living donor nephrectomy, will be randomized into a group with deep or moderate neuromuscular blockade. Deep neuromuscular blockade is defined as post tetanic count 1-2.

Main study parameters/endpoints: The primary outcome measurement will be the Quality of Recovery-40 questionnaire (overall score) at 48 hours after extubation.

Secondary outcomes measured are: intra-operative parameters (e.g. surgical conditions, operation time, length of pneumoperitoneum, first warm ischemia time, estimated blood loss, conversion to open or hand-assisted donor nephrectomy, intra-operative complications, cumulative use of rocuronium and sugammadex), the total score of the quality of Recovery-40 questionnaire at 48 hours after extubation, post-operative pain (components of pain scores); postoperative nausea and vomiting (NRS), the cumulative use of analgesics and anti-emetics, time to reach discharge criteria and postoperative complications.

ELIGIBILITY:
All adult individuals, who are scheduled for living kidney donation.

Inclusion Criteria:

* obtained informed consent
* age over 18 years

Exclusion Criteria:

* insufficient control of the Dutch language to read the patient information and to fill out the questionnaires
* chronic use of analgesics or psychotropic drugs
* use of NSAIDs shorter than 5 days before surgery
* known or suspect allergy to rocuronium of sugammadex
* neuromuscular disease
* indication for rapid sequence induction
* deficiency of vitamin K-dependent clotting factors, coagulopathy or active use of coumarin derivates.
* Peri-operative use of fusidic acid or flucloxacillin
* Severe renal impairment (creatinine clearance <30ml/min)
* Morbid obesity (BMI>35 kg/m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moira Bruintjes, Msc., Principal Investigator — Radboud University Medical Center; Michiel Warlé, Dr., Principal Investigator — Radboud University Medical Center; Andries E Braat, Dr., Principal Investigator — LUMC
Locations (2):
- Netherlands (2):
  - LUMC, Leiden
  - Radboudumc, Nijmegen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reijnders-Boerboom GTJA, van Helden EV, Minnee RC, Albers KI, Bruintjes MHD, Dahan A, Martini CH, d'Ancona FCH, Scheffer GJ, Keijzer C, Warle MC. Deep neuromuscular block reduces the incidence of intra-operative complications during laparoscopic donor nephrectomy: a pooled analysis of randomized controlled trials. Perioper Med (Lond). 2021 Dec 9;10(1):56. doi: 10.1186/s13741-021-00224-1. PMID 34879862
- [Derived] Albers KI, van Helden EV, Dahan A, Martini CH, Bruintjes MHD, Scheffer GJ, Steegers MAH, Keijzer C, Warle MC. Early postoperative pain after laparoscopic donor nephrectomy predicts 30-day postoperative infectious complications: a pooled analysis of randomized controlled trials. Pain. 2020 Jul;161(7):1565-1570. doi: 10.1097/j.pain.0000000000001842. PMID 32107359
- [Derived] Bruintjes MHD, Krijtenburg P, Martini CH, Poyck PP, d'Ancona FCH, Huurman VAL, van der Jagt M, Langenhuijsen JF, Nijboer WN, van Laarhoven CJHM, Dahan A, Warle MC; RELAX collaborator group. Efficacy of profound versus moderate neuromuscular blockade in enhancing postoperative recovery after laparoscopic donor nephrectomy: A randomised controlled trial. Eur J Anaesthesiol. 2019 Jul;36(7):494-501. doi: 10.1097/EJA.0000000000000992. PMID 30920983
- [Derived] Bruintjes MH, Braat AE, Dahan A, Scheffer GJ, Hilbrands LB, d'Ancona FC, Donders RA, van Laarhoven CJ, Warle MC. Effectiveness of deep versus moderate muscle relaxation during laparoscopic donor nephrectomy in enhancing postoperative recovery: study protocol for a randomized controlled study. Trials. 2017 Mar 4;18(1):99. doi: 10.1186/s13063-017-1785-y. PMID 28259181

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 26 patients were assessed for eligibility but excluded, 8 patients did not meet the inclusion criteria 18 patients declined to participate
Period: Overall Study
Arm/Group | Group A: Deep Neuromuscular Blockade | Group B: Moderate Neuromuscular Blockade
Started | 50 | 51
Completed | 48 | 48
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — logistic problems | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group A: Deep Neuromuscular Blockade: An extra bolus of rocuronium after intubation followed by infusion
  Rocuronium: A bolus of 0.7 mg/kg rocuronium is administered just after tracheal intubation and then an infusion of rocuronium (0.3 to 0.4 mg/kg) is started when PTC is more than 0 and titrated towards PTC 1-2.
- Total: Total of all reporting groups
Arm/Group | Group A: Deep Neuromuscular Blockade | Group B: Moderate Neuromuscular Blockade | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (10.2) | 56.6 (9.7) | 56.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Distribution of participants per sex
  Participants
    Female | 27 | 24 | 51
    Male | 21 | 24 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m2] | 26.7 (2.9) | 26.5 (3.0) | 26.6 (3.0)
Centre [Count of Participants; unit: Participants] — Distribution of participants per centre
  Participants
    Radboud | 35 | 38 | 73
    LUMC | 13 | 10 | 23
Previous abdominal surgery [Count of Participants; unit: Participants] — Number of participants with previous abdominal surgery
  Participants | 13 | 10 | 23
Previous pregnancies [Count of Participants; unit: Participants] — Number of participants with previous pregnancies
  Participants | 21 | 21 | 42
Side of nephrectomy [Count of Participants; unit: Participants] — Distribution of participants per side of nephrectomy
  Participants
    Left | 42 | 42 | 84
    Right | 6 | 6 | 12
Vascular anatomy (more than one renel artery or renal vein) [Count of Participants; unit: Participants] — Number of participants with more than one renal artery or renal vein
  Participants | 13 | 17 | 30

OUTCOME MEASURES:

1. Primary Outcome: Total Score of the Quality of Recovery-40 Questionnaire (QoR-40)
Description: The QoR-40 is a validated assessment tool for measuring a patient's self-assessed quality of recovery after surgery. It consists of 40 questions measuring 5 dimensions: patient support, comfort, emotions, physical independence and pain. Each item is rated on a scale of 1 to 5, giving a minimal score of 40 and a maximum score of 200. Higher values represent a better outcome
Time Frame: Day 1: 24 hours after detubation
Population: Explanation of missing data:
  One patient from group A missed one page of the QOR-40 questionnaire on postoperative day 1.
  One patient from group B did not complete the questionnaires on postoperative days 1 and 2 because of personal circumstances
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A: Deep Neuromuscular Blockade | Group B: Moderate Neuromuscular Blockade
Number analyzed (Participants) | 47 | 47
score on a scale | 169.3 (18.3) | 169.5 (15.5)

2. Secondary Outcome: Surgical Conditions
Description: Surgical rating score, concerning the quality of the surgical field, scored with the surgical rating scale (SRS) A likert scale from 1 to 5. Higher scores represent better outcomes.
  1. = extremely poor conditions
  2. = poor conditions
  3. = acceptable conditions
  4. =good conditions
  5. = optimal conditions
Time Frame: Day 0: Intraoperative, average of scores up to 240 minutes (assessed each 15 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A: Deep Neuromuscular Blockade | Group B: Moderate Neuromuscular Blockade
Number analyzed (Participants) | 48 | 48
score on a scale | 4.8 (0.3) | 4.7 (0.5)

3. Secondary Outcome: Length of Pneumoperitoneum
Description: Intraoperative parameter of duration of pneumoperitoneum
Time Frame: Day 0: once, up to 240 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group A: Deep Neuromuscular Blockade | Group B: Moderate Neuromuscular Blockade
Number analyzed (Participants) | 48 | 48
minutes | 122.8 (44.5) | 113.8 (39.2)

4. Secondary Outcome: Warm Ischemia Time
Description: Intraoperative parameter measuring the time (in minutes) between dissection of the renal artery and flushing of the kidney after retrieval
Time Frame: Day 0: once, up to 240 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group A: Deep Neuromuscular Blockade | Group B: Moderate Neuromuscular Blockade
Number analyzed (Participants) | 48 | 48
minutes | 3.6 (1.3) | 3.9 (1.6)

5. Secondary Outcome: Estimated Blood Loss
Description: Intraoperative parameter
Time Frame: Day 0: once, up to 240 minutes
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Group A: Deep Neuromuscular Blockade | Group B: Moderate Neuromuscular Blockade
Number analyzed (Participants) | 48 | 48
ml | 60.2 (68.5) | 69.1 (72.3)

6. Secondary Outcome: Conversion
Description: Number of Participants with conversion to open or hand-assisted donor nephrectomy
Time Frame: Day 0: once, up to 240 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Deep Neuromuscular Blockade | Group B: Moderate Neuromuscular Blockade
Number analyzed (Participants) | 48 | 48
Participants | 0 | 2

7. Secondary Outcome: Intra-operative Complications
Description: Number of Participants with Complications which occurred during surgery
Time Frame: Day 0: once, up to 240 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Deep Neuromuscular Blockade | Group B: Moderate Neuromuscular Blockade
Number analyzed (Participants) | 48 | 48
Participants | 1 | 6

8. Secondary Outcome: Cumulative Use of Rocuronium
Description: Total amount of rocuronium administered during surgery
Time Frame: Day 0: once, up to 240 minutes
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Group A: Deep Neuromuscular Blockade | Group B: Moderate Neuromuscular Blockade
Number analyzed (Participants) | 48 | 48
mg | 184.6 (83.1) | 67.0 (41.2)

9. Secondary Outcome: Total Score of the Quality of Recovery-40 Questionnaire
Description: as for outcome 1
Time Frame: Day 2: 48 hours after detubation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A: Deep Neuromuscular Blockade | Group B: Moderate Neuromuscular Blockade
Number analyzed (Participants) | 48 | 47
score on a scale | 175.6 (17.8) | 175.3 (16.5)

10. Secondary Outcome: Postoperative Pain
Description: components of pain scores after 1 hour, 6 hours, on postoperative day 1 (POD1) and postoperative day 2 (POD2).
  Likert scale from 0 to 10. Higher scores represent more pain.
Time Frame: Day 0: 1h, 6h, day 1: 24h and day 2: 48 hours (and if still admitted 72h) after detubation
Population: 1 patient from the moderate NMB group was not able to complete the questionnaires on day 1 and day 2 because of personal circumstances.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A: Deep Neuromuscular Blockade | Group B: Moderate Neuromuscular Blockade
Number analyzed (Participants) | 48 | 48
score on a scale
  Overall_1h (PACU) | 4.0 (2.3) | 4.31 (2.4)
  Referred pain_1h (PACU) | 0.0 (0.2) | 0.3 (1.1)
  overall_6h | 3.7 (2.7) | 4.5 (2.2)
  Referred pain_6h | 0.7 (1.6) | 1.0 (1.8)
  Overall_POD1: number analyzed (Participants) | 48 | 47
  Overall_POD1 | 5.0 (2.3) | 5.6 (2.1)
  Referred pain+POD1: number analyzed (Participants) | 48 | 47
  Referred pain+POD1 | 2.5 (2.7) | 3.2 (2.8)
  Overall_POD2: number analyzed (Participants) | 48 | 47
  Overall_POD2 | 4.6 (1.9) | 4.9 (2.2)
  Referred pain_POD2: number analyzed (Participants) | 48 | 47
  Referred pain_POD2 | 2.4 (2.7) | 3.3 (2.9)

11. Secondary Outcome: Postoperative Complications
Description: Number of participants with postoperative complications that occurred up to 8 weeks after surgery
Time Frame: 24 and 48 hours (and if still admitted 72h) after detubation and 4 and 8 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Deep Neuromuscular Blockade | Group B: Moderate Neuromuscular Blockade
Number analyzed (Participants) | 48 | 48
Participants
  during hospital stay | 2 | 4
  30 days after surgery | 7 | 5
  60 days after surgery | 9 | 5

12. Secondary Outcome: Discharge Criteria
Description: Scoring the following criteria: adequate pain control with oral medication, passage of flatus or defecation, intake of solid food tolerated, patient is mobilized and independent and patient accepts discharge.
Time Frame: 24 and 48 hours after detubation
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Deep Neuromuscular Blockade | Group B: Moderate Neuromuscular Blockade
Number analyzed (Participants) | 48 | 48
Participants
  reached all criteria after 24hours | 13 | 15
  reached all criteria after 48 hours | 24 | 29

13. Secondary Outcome: Pain Scores
Description: Total amount of pain 4 weeks after surgery Likert scale from 0 to 10. Higher scores represent more pain (worse outcome).
Time Frame: once, 4 weeks after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A: Deep Neuromuscular Blockade | Group B: Moderate Neuromuscular Blockade
Number analyzed (Participants) | 48 | 48
score on a scale | 1.88 (1.91) | 1.85 (1.92)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Group A: Deep Neuromuscular Blockade | Group B: Moderate Neuromuscular Blockade
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 1/48
Other Adverse Events (participants affected / at risk) | 9/48 | 5/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Deep Neuromuscular Blockade (N=48) | Group B: Moderate Neuromuscular Blockade (N=48)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Deep Neuromuscular Blockade (N=48) | Group B: Moderate Neuromuscular Blockade (N=48)
Urinary tract infection (Infections and infestations) | 6 (6) | 4 (4)
Wound infection (Infections and infestations) | 2 (2) | 0 (0)
Hypertension (General disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
It appeared to be difficult to achieve and maintain the intended depth of neuromuscular blockade. Despite high dosages of rocuronium with continuous infusion, the intended deep NMB was not achieved in all patients within the deep NMB group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT02838134/Prot_SAP_000.pdf